CLINICAL TRIAL: NCT06112366
Title: Comparison of the Efficiency of Tissue Adhesive (Periacryl 90) and Silk Suture in Bilateral Mandibular Impacted Wisdom Teeth Surgery
Brief Title: Comparison of Silk Suture and Tissue Adhesive for Wound Closure After Impacted Tooth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Serap Keskin Tunc, Associate Professor Serap Keskin Tunc, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: YYU-04/05.18.2022
Record Dates: First submitted 2023-10-17; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Tooth, Impacted; Tooth Diseases
Keywords: impacted wisdom teeth; tissue adhesive; silk suture
MeSH Terms: conditions — Tooth, Impacted; Tooth Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group used tissue adhesive for wound closure after extraction of impacted wisdom teeth (Experimental): In this study of 30 patients, 21 females and 9 males, 60 fully impacted lower wisdom teeth were extracted bilaterally and in the same position. One of the bilaretal teeth of the patients was randomly selected and tissue adhesive (Periacryl 90) was applied for wound closure as an experimental group.
  Interventions: Procedure: Surgery of impacted mandibular wisdom teeth
- Control group used silk sutures after extraction of impacted wisdom teeth (Placebo Comparator): Bilateral impacted wisdom teeth of the patients were randomly selected. After the tooth in the experimental group was extracted, the other impacted wisdom tooth was selected as the control group and silk sutures were used for wound closure.
  Interventions: Procedure: Surgery of impacted mandibular wisdom teeth (the other side)

INTERVENTIONS:
Procedure: Surgery of impacted mandibular wisdom teeth — All surgical procedures were performed by the same surgeon using the standard surgical technique described below. The anesthetic used was 4% articaine with 1:100,000 adrenaline. In all patients, a sulcus incision was made in the lower second molar and an envelope incision in the third molar region, the mucoperiosteal flap was removed, and extraction was performed with a bone elevator and a third molar elevator. If necessary, the impacted molar was incised with a high-speed dental handpiece and a fissure bur. The wound was irrigated with saline and the wound edges were sealed with tissue adhesive containing cyanoacrylate.
  Other Names: Surgery of impacted molar teeth
  Arms: The study group used tissue adhesive for wound closure after extraction of impacted wisdom teeth
Procedure: Surgery of impacted mandibular wisdom teeth (the other side) — All surgical procedures were performed by the same surgeon using the standard surgical technique described below. The anesthetic used was 4% articaine with 1:100,000 adrenaline. In all patients, a sulcus incision was made in the lower second molar and an envelope incision in the third molar region, the mucoperiosteal flap was removed, and extraction was performed with a bone elevator and a third molar elevator. If necessary, the impacted molar was incised with a high-speed dental handpiece and a fissure bur. The wound was irrigated with copious amounts of saline, and the wound edges were carefully sutured with simple 4.0 silk braided non-absorbable sutures.
  Other Names: Surgery of impacted molar teeth
  Arms: Control group used silk sutures after extraction of impacted wisdom teeth

SUMMARY:
This study was administered to 21 female and 9 male patients. Patients with impacted wisdom teeth on both sides of the mandible were selected. After extraction of the impacted teeth, silk sutures were used on one side and cyanoacrylate tissue adhesive on the other side for wound closure. The effects of these two materials on patient comfort were investigated.

DETAILED DESCRIPTION:
The aim of this study was to compare the effectiveness of tissue adhesive (Periacryl 90) and silk suture in bilateral mandibular impacted wisdom tooth surgery. In the study of 30 patients, 21 females and 9 males, 60 fully impacted lower wisdom teeth were extracted bilaterally and in the same position. One of the bilaretal teeth of the patients was randomly selected and tissue adhesive (Periacryl 90) was applied for wound closure as the experimental group, while the other tooth was selected as the control group and the wound was closed with silk suture. The selected side was determined by a closed envelope procedure. After the first impacted tooth extraction, the patient waited until the wound healed and the symptoms disappeared completely, and then the other tooth was extracted. Both extractions were evaluated on days 3 and 7 for wound healing, edema and trismus. Wound healing was evaluated as good, acceptable and poor. VAS (Visual Analog Scale) was used for pain assessment

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with bilateral fully impacted mandibular wisdom teeth

Exclusion Criteria:

* Patients were excluded from the study if they did not understand the clinical procedures of the study,
* Had allergies or intolerance to any of the substances used in the study,
* Patients on anticoagulant or psychiatric treatment,
* Pregnant or breastfeeding,
* Patients using oral contraceptiveswere,
* Diabetic,
* Patients with periodontal disease or active infection,
* Poor oral hygiene

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Mouth opening measurements | 0-28 days
  The distance between the incisals of the patient's central teeth at maximal mouth opening.
Facial edema | 0-28 days
  Measurement between facial craniometric points (angulus-tragus, angulus-lateral canthus, angulus-nasal base, angulus-lateral canthus, and angulus-pogonion). The number of participants in the split mouth model was 22. A total of 44 impacted teeth were extracted and edema was measured before and 1 week after each extraction.
Wound healing | 0-28 days
  View of the wound site in the operation area. The REEDA scale was used for the clinical evaluation of the intraoral surgical field. This scale It includes five factors that indicate wound healing: Redness, Edema, Echymosis, Discharge, Approximation. Each of the recovery factors is evaluated by giving scores of 0, 1, 2 and 3 and the sum of the scores obtained as a result of the evaluation of these five categories constitutes the REEDA score. The lowest score is 0 and the highest score is 15.
Visual Analog Scale | 0-28 days
  A numerical rating scale VAS was used for pain analysis (0=no pain, 10=most severe pain). The pain levels at 24 hours, 48 hours and 1 week after the surgical procedure were recorded on the patient follow-up form by all patients who participated in the study by explaining that there was no pain at the "zero" level and the most severe pain known at the "10" level on the pain scale, which was organized as a 10 cm horizontal line on the prepared forms.

CONTACTS AND LOCATIONS:
Locations (1):
- Serap Keskin Tunc, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided